CLINICAL TRIAL: NCT06055192
Title: Prevalence and Burden of Nausea and Vomiting in Pregnant Women in Switzerland: Survey Purity 2022
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Effik SA (Other)
Collaborators: Opera CRO, a TIGERMED Group Company (Other)
Responsible Party: Sponsor
Other Study IDs: OPEFF/0122/SU
Record Dates: First submitted 2023-09-20; First posted 2023-09-26 (Actual); Last update posted 2023-09-26 (Actual); Status verified 2023-09

CONDITIONS: Nausea; Vomiting of Pregnancy
Keywords: Nausea; Vomiting; Pregnancy
MeSH Terms: conditions — Nausea; Vomiting | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Survey — Survey

SUMMARY:
The latest data on the prevalence of nausea in pregnancy in Switzerland is dated 2015 but has been hypothesised that the recent introduction on the market of new drugs against this symptom could modify its epidemiology. For this reason, we have planned the present survey, calculating an adequate sample size of Swiss pregnant women (the population of interest) and, according to a cross-sectional design, planning the collection of response variables with the aim of estimating the prevalence of burden and nausea and vomiting in pregnancy

DETAILED DESCRIPTION:
Nausea with or without vomiting (Nausea and Vomiting in Pregnancy - NVP) in early pregnancy (before 9 and up to 16 weeks of gestation) is very common (50-80%); these symptoms rarely persist throughout pregnancy (10-20%). Even if NVP aetiology remains unknown, the cause is most likely multifactorial NVP severity can be assessed with the validated, 24-hour Pregnancy-Unique Quantification of Emesis (PUQE-24) Scale.

Management and treatment of NVP focus on reducing symptoms, improving quality of life, preventing serious complications, and minimising foetal effects of maternal pharmacologic treatment. It is advised to follow dietary and lifestyle recommendations, followed by available alternative and pharmacological treatments.

Swissmedic has recently approved doxylamine as a drug for the treatment of NVP symptoms in combination with pyridoxine (Cariban®, Effik SA, Switzerland). Its efficacy and safety have been widely studied. A 2014 data re-analysis of a previous meta-analysis took into account a total of 139414 women in reports about the safety of antihistamines and 129108 in reports about the safety of doxylamine. In these studies, 23485 women were exposed to antihistamines and 14624 were exposed to doxylamine. Neither increased foetal risk for congenital malformations nor other adverse pregnancy outcomes were demonstrated. The safety of the drug is additionally supported by extensive international literature.

Moreover, a recent study showed that Cariban® behaves as a prolonged-release formulation, which correlates with rapid absorption and arising of the actives in the plasma, but also long-lasting and sustained bioavailability, especially when administered following the complete posology. These results would underlie its demonstrated efficacy to relieve nausea and vomiting of pregnancy (NVP) under clinical settings.

The exposure to doxylamine-pyridoxine in pregnancy (or to the combination of doxylamine and pyridoxine) is classified as safe, and its use is recommended as first-line therapy of nausea and vomiting in pregnancy by the American College of Obstetricians and Gynaecologists (ACOG) Guidelines, by the Society of Obstetricians and Gynecologists of Canada and organizations such as Mother to Baby (formerly known as Organization of Teratogen Information Services.

An epidemiological study, published in 2015, stated that the prevalence of nausea in Switzerland was 70,6%. It is to be noted that women who reported nausea also had a high burden of co-morbidity, especially heartburn and reflux symptoms and an association of NPV with symptoms of depression and sick leave was shown.

It is possible that the recent introduction of an association of doxylamine succinate 10 mg and pyridoxine hydrochloride 10 mg (Cariban®, Effik SA Switzerland) on the Swiss market and the recent publication of the SGGG Expert letter on NVP and hyperemesis gravidarum (1) could have had a substantial impact on the extent of this disturbance, the awareness of the therapists and the perception of the women.

In this context, a Survey will be carried out. A Survey is a procedure which, through a scientific method of detection (a questionnaire to be submitted to a representative sample of subjects related to the issue of the research) allows to collect, and subsequently to analyse, the data to study the relationships between different variables would yield significant scientific results.

The objectives of the study are: Evaluate the prevalence and burden that the symptoms of nausea and vomiting have in pregnant women in Switzerland.

The following outcomes will be evaluated:

* Demographic data (including ethnicity: Caucasian, African, Asian, or Other).
* NVP prevalence.
* Percentage of mild, medium, and severe cases based on PUQE-24.
* Percentage of answer allocation to NVP related questions.
* Onset for each symptom and its duration.
* Correlations between demographic data (age, first pregnancy status, multiparity, geographical origin, kinds of work and educational qualification) and the presence of symptoms and their severity.
* Correlation of the above-mentioned parameters with the use of non-pharmacological, pharmacological or both therapies.
* Analysis of drug therapies, of their correlation with the severity of the symptoms during pregnancy and with the possible outcomes of the same.
* Correlation between the severity of the symptoms and the consequences on the woman's personal life (family, work, etc.).
* Number of cases with hospitalization in relation to total and severity of symptoms (PUQE-24).
* Correlation between symptoms in pregnancy and outcomes based on data from the post pregnancy questionnaire (weight of the new-born, gestational age at birth and any complications).

ELIGIBILITY:
Inclusion Criteria:

Subjects will be eligible for inclusion if all the following criteria are respected:

* Women aged ≥ 18 years.
* Women in physiological pregnancy and between the 18th and 22nd week of pregnancy (at time of morphological ultrasound).
* Women able to communicate adequately with the Investigator and able to read, understand and provide the answers required by the questionnaires in one of the languages in which they will be provided (Italian, German, French or English).
* Women able to understand and who can provide valid informed consent to the Survey.

Exclusion Criteria:

* Subjects fulfilling one or more of the following exclusion criteria will not be included in the study:

  * Twin pregnancy.
  * Medically assisted procreation (MAP).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — 200 women during the weeks 18-22 of their pregnancy
Study Population: 200 women during the weeks 18-22 of their pregnancy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2023-09 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-10 (Estimated)

PRIMARY OUTCOMES:
Primary Outcome Measure | 185 days
  Evaluate the prevalence and burden that the symptoms of nausea and vomiting have in pregnant women in Switzerland

SECONDARY OUTCOMES:
Secondary Outcome Measure | 185 days
  demographic data (including ethnicity: Caucasian, African, Asian or Other).
Secondary Outcome Measure | 185 days
  NVP prevalence
Secondary Outcome Measure | 185 days
  Percentage of mild, medium, and severe cases based on PUQE-24.
Secondary Outcome Measure | 185 days
  Percentage of answer allocation to NVP related questions
Secondary Outcome Measure | 185 days
  Onset for each symptom and its duration
Secondary Outcome Measure | 185 days
  Correlations between demographic data (age, first pregnancy status, multiparity, geographical origin, kinds of work and educational qualification) and the presence of symptoms and their severity.
Secondary Outcome Measure | 185 days
  Correlation of the above-mentioned parameters with the use of non-pharmacological, pharmacological (e.g., Cariban®) or both therapies.
Secondary Outcome Measure | 185 days
  Analysis of drug therapies, their correlation with the severity of the symptoms during pregnancy and with the possible outcomes of the same
Secondary Outcome Measure | 185 days
  Correlation between the severity of the symptoms and the consequences on the woman's personal life (family, work, etc.).
Secondary Outcome Measure | 185 days
  Number of cases with hospitalization in relation to total and severity of symptoms (PUQE-24).
Secondary Outcome Measure | 185 days
  Correlation between symptoms in pregnancy and outcomes based on data from the post pregnancy questionnaire (weight of the new-born, gestational age at birth and any complications).

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] SR 810.301 - Ordinance of 20 September 2013 on Human Research with the Exception of Clinical Trials (Human Research Ordinance, HRO) [Internet]. [cited 2022 Jun 13]. Available from: https://www.fedlex.admin.ch/eli/cc/2013/642/en
- [Background] fedlex-data-admin-ch-eli-cc-2013-643-20140101-en-pdf-a.pdf [Internet]. [cited 2022 Jun 13]. Available from: https://fedlex.data.admin.ch/filestore/fedlex.data.admin.ch/eli/cc/2013/643/20140101/en/pdf-a/fedlex-data-admin-ch-eli-cc-2013-643-20140101-en-pdf-a.pdf
- [Background] WMA - The World Medical Association-WMA Declaration of Helsinki - Ethical Principles for Medical Research Involving Human Subjects [Internet]. [cited 2022 Jun 13]. Available from: https://www.wma.net/policies-post/wma-declaration-of-helsinki-ethical-principles-for-medical-research-involving-human-subjects/
- [Background] Martinez de Tejada B, Vonzun L, Von Mandach DU, Burch A, Yaron M, Hodel M, Surbek D, Hoesli I. Nausea and vomiting of pregnancy, hyperemesis gravidarum. Eur J Obstet Gynecol Reprod Biol. 2025 Jan;304:115-120. doi: 10.1016/j.ejogrb.2024.11.006. Epub 2024 Nov 5. No abstract available. PMID 39612885
- [Background] Ebrahimi N, Maltepe C, Bournissen FG, Koren G. Nausea and vomiting of pregnancy: using the 24-hour Pregnancy-Unique Quantification of Emesis (PUQE-24) scale. J Obstet Gynaecol Can. 2009 Sep;31(9):803-807. doi: 10.1016/S1701-2163(16)34298-0. PMID 19941704
- [Background] Koren G, Boskovic R, Hard M, Maltepe C, Navioz Y, Einarson A. Motherisk-PUQE (pregnancy-unique quantification of emesis and nausea) scoring system for nausea and vomiting of pregnancy. Am J Obstet Gynecol. 2002 May;186(5 Suppl Understanding):S228-31. doi: 10.1067/mob.2002.123054. PMID 12011891
- [Background] Koren G, Cohen R. Measuring the severity of nausea and vomiting of pregnancy; a 20-year perspective on the use of the pregnancy-unique quantification of emesis (PUQE). J Obstet Gynaecol. 2021 Apr;41(3):335-339. doi: 10.1080/01443615.2020.1787968. Epub 2020 Aug 19. PMID 32811235
- [Background] Lee NM, Saha S. Nausea and vomiting of pregnancy. Gastroenterol Clin North Am. 2011 Jun;40(2):309-34, vii. doi: 10.1016/j.gtc.2011.03.009. PMID 21601782
- [Background] McParlin C, O'Donnell A, Robson SC, Beyer F, Moloney E, Bryant A, Bradley J, Muirhead CR, Nelson-Piercy C, Newbury-Birch D, Norman J, Shaw C, Simpson E, Swallow B, Yates L, Vale L. Treatments for Hyperemesis Gravidarum and Nausea and Vomiting in Pregnancy: A Systematic Review. JAMA. 2016 Oct 4;316(13):1392-1401. doi: 10.1001/jama.2016.14337. PMID 27701665
- [Background] Nuangchamnong N, Niebyl J. Doxylamine succinate-pyridoxine hydrochloride (Diclegis) for the management of nausea and vomiting in pregnancy: an overview. Int J Womens Health. 2014 Apr 12;6:401-9. doi: 10.2147/IJWH.S46653. eCollection 2014. PMID 24748822
- [Background] Madjunkova S, Maltepe C, Koren G. The delayed-release combination of doxylamine and pyridoxine (Diclegis(R)/Diclectin (R)) for the treatment of nausea and vomiting of pregnancy. Paediatr Drugs. 2014 Jun;16(3):199-211. doi: 10.1007/s40272-014-0065-5. PMID 24574047
- [Background] Gilboa SM, Ailes EC, Rai RP, Anderson JA, Honein MA. Antihistamines and birth defects: a systematic review of the literature. Expert Opin Drug Saf. 2014 Dec;13(12):1667-98. doi: 10.1517/14740338.2014.970164. Epub 2014 Oct 11. PMID 25307228
- [Background] Einarson TR, Leeder JS, Koren G. A method for meta-analysis of epidemiological studies. Drug Intell Clin Pharm. 1988 Oct;22(10):813-24. doi: 10.1177/106002808802201021. PMID 3229352
- [Background] McKeigue PM, Lamm SH, Linn S, Kutcher JS. Bendectin and birth defects: I. A meta-analysis of the epidemiologic studies. Teratology. 1994 Jul;50(1):27-37. doi: 10.1002/tera.1420500105. PMID 7974252
- [Background] Koren G, Clark S, Hankins GD, Caritis SN, Miodovnik M, Umans JG, Mattison DR. Effectiveness of delayed-release doxylamine and pyridoxine for nausea and vomiting of pregnancy: a randomized placebo controlled trial. Am J Obstet Gynecol. 2010 Dec;203(6):571.e1-7. doi: 10.1016/j.ajog.2010.07.030. Epub 2010 Sep 16. PMID 20843504
- [Background] Chin JW, Gregor S, Persaud N. Re-analysis of safety data supporting doxylamine use for nausea and vomiting of pregnancy. Am J Perinatol. 2014 Sep;31(8):701-10. doi: 10.1055/s-0033-1358772. Epub 2013 Dec 9. PMID 24323370
- [Background] Seto A, Einarson T, Koren G. Pregnancy outcome following first trimester exposure to antihistamines: meta-analysis. Am J Perinatol. 1997 Mar;14(3):119-24. doi: 10.1055/s-2007-994110. PMID 9259911
- [Background] Lee J, Einarson A, Gallo M, Okotore B, Koren G. Longitudinal change in the treatment of nausea and vomiting of pregnancy in Ontario. Can J Clin Pharmacol. 2000 Winter;7(4):205-8. PMID 11118967
- [Background] Persaud N, Chin J, Walker M. Should doxylamine-pyridoxine be used for nausea and vomiting of pregnancy? J Obstet Gynaecol Can. 2014 Apr;36(4):343-348. doi: 10.1016/S1701-2163(15)30611-3. PMID 24798673
- [Background] Smolina K, Hanley GE, Mintzes B, Oberlander TF, Morgan S. Trends and Determinants of Prescription Drug Use during Pregnancy and Postpartum in British Columbia, 2002-2011: A Population-Based Cohort Study. PLoS One. 2015 May 26;10(5):e0128312. doi: 10.1371/journal.pone.0128312. eCollection 2015. PMID 26011706
- [Background] Koren G. Safety considerations surrounding use of treatment options for nausea and vomiting in pregnancy. Expert Opin Drug Saf. 2017 Nov;16(11):1227-1234. doi: 10.1080/14740338.2017.1361403. Epub 2017 Aug 9. PMID 28749713
- [Background] Fejzo MS, Trovik J, Grooten IJ, Sridharan K, Roseboom TJ, Vikanes A, Painter RC, Mullin PM. Nausea and vomiting of pregnancy and hyperemesis gravidarum. Nat Rev Dis Primers. 2019 Sep 12;5(1):62. doi: 10.1038/s41572-019-0110-3. PMID 31515515
- [Background] Doxylamine/pyridoxine for nausea and vomiting in pregnancy. Drug Ther Bull. 2019 Mar;57(3):38-41. doi: 10.1136/dtb.2018.000053. Epub 2019 Jan 31. No abstract available. PMID 30705026
- [Background] Brott NR, Reddivari AKR. Doxylamine. In: StatPearls [Internet]. Treasure Island (FL): StatPearls Publishing; 2023 [cited 2023 Jun 22]. Available from: http://www.ncbi.nlm.nih.gov/books/NBK551646/
- [Background] Biffi A, Rea F, Locatelli A, Cetin I, Filippelli A, Corrao G. Misleading meta-analyses of observational studies may generate unjustified alarms: The case of medications for nausea and vomiting in pregnancy. Pharmacol Res. 2021 Jan;163:105229. doi: 10.1016/j.phrs.2020.105229. Epub 2020 Oct 5. PMID 33031909
- [Background] Berard A, Sheehy O, Gorgui J, Zhao JP, Soares de Moura C, Bernatsky S. New evidence for concern over the risk of birth defects from medications for nausea and vomitting of pregnancy. J Clin Epidemiol. 2019 Dec;116:39-48. doi: 10.1016/j.jclinepi.2019.07.014. Epub 2019 Jul 26. PMID 31352006
- [Background] Brent RL. Bendectin: review of the medical literature of a comprehensively studied human nonteratogen and the most prevalent tortogen-litigen. Reprod Toxicol. 1995 Jul-Aug;9(4):337-49. doi: 10.1016/0890-6238(95)00020-b. PMID 7496090
- [Background] Neutel CI, Johansen HL. Measuring drug effectiveness by default: the case of Bendectin. Can J Public Health. 1995 Jan-Feb;86(1):66-70. PMID 7728721
- [Background] Saz-Leal P, Zamorano-Dominguez L, Frias J, Guerra P, Saura-Valls M, Roca-Juanes R, Nebot-Troyano J, Garcia-Aguilar E, Vilchez T, Urso K. Bioavailability of Cariban(R) Capsules: A Modified-Release Fixed-Dose Combination of Doxylamine and Pyridoxine to Relieve Nausea and Vomiting During Pregnancy. Drugs R D. 2023 Jun;23(2):185-195. doi: 10.1007/s40268-023-00425-7. Epub 2023 Jun 15. PMID 37318714
- [Background] London V, Grube S, Sherer DM, Abulafia O. Hyperemesis Gravidarum: A Review of Recent Literature. Pharmacology. 2017;100(3-4):161-171. doi: 10.1159/000477853. Epub 2017 Jun 23. PMID 28641304
- [Background] Committee on Practice Bulletins-Obstetrics. ACOG Practice Bulletin No. 189: Nausea And Vomiting Of Pregnancy. Obstet Gynecol. 2018 Jan;131(1):e15-e30. doi: 10.1097/AOG.0000000000002456. PMID 29266076
- [Background] APGO. APGO. Nausea and vomiting of pregnancy. APGO Educational series on women's health issues. Boston: Jespersen & Associates, LLC; 2013. 2013.
- [Background] Arsenault MY, Lane CA, MacKinnon CJ, Bartellas E, Cargill YM, Klein MC, Martel MJ, Sprague AE, Wilson AK. The management of nausea and vomiting of pregnancy. J Obstet Gynaecol Can. 2002 Oct;24(10):817-31; quiz 832-3. English, French. PMID 12405123
- [Background] Nausea and Vomiting of Pregnancy (NVP). 2022;
- [Background] Madjunkova S, Maltepe C, Koren G. The Leading Concerns of American Women with Nausea and Vomiting of Pregnancy Calling Motherisk NVP Helpline. Obstet Gynecol Int. 2013;2013:752980. doi: 10.1155/2013/752980. Epub 2013 Apr 15. PMID 23690784
- [Background] Heitmann K, Solheimsnes A, Havnen GC, Nordeng H, Holst L. Treatment of nausea and vomiting during pregnancy -a cross-sectional study among 712 Norwegian women. Eur J Clin Pharmacol. 2016 May;72(5):593-604. doi: 10.1007/s00228-016-2012-6. Epub 2016 Jan 27. PMID 26815908
- [Background] Heitmann K, Holst L, Lupattelli A, Maltepe C, Nordeng H. Treatment of nausea in pregnancy: a cross-sectional multinational web-based study of pregnant women and new mothers. BMC Pregnancy Childbirth. 2015 Dec 1;15:321. doi: 10.1186/s12884-015-0746-2. PMID 26628289
- [Background] Heitmann K, Nordeng H, Havnen GC, Solheimsnes A, Holst L. The burden of nausea and vomiting during pregnancy: severe impacts on quality of life, daily life functioning and willingness to become pregnant again - results from a cross-sectional study. BMC Pregnancy Childbirth. 2017 Feb 28;17(1):75. doi: 10.1186/s12884-017-1249-0. PMID 28241811
- [Background] Rubenfeld GD. Surveys: an introduction. Respir Care. 2004 Oct;49(10):1181-5. PMID 15447800
- [Background] Safdar N, Abbo LM, Knobloch MJ, Seo SK. Research Methods in Healthcare Epidemiology: Survey and Qualitative Research. Infect Control Hosp Epidemiol. 2016 Nov;37(11):1272-1277. doi: 10.1017/ice.2016.171. Epub 2016 Aug 12. PMID 27514583
- [Background] von Elm E, Altman DG, Egger M, Pocock SJ, Gotzsche PC, Vandenbroucke JP; STROBE Initiative. The Strengthening the Reporting of Observational Studies in Epidemiology (STROBE) statement: guidelines for reporting observational studies. J Clin Epidemiol. 2008 Apr;61(4):344-9. doi: 10.1016/j.jclinepi.2007.11.008. PMID 18313558
- [Background] Office FS. Births [Internet]. [cited 2022 Jun 14]. Available from: https://www.bfs.admin.ch/bfs/en/home/statistiken/bevoelkerung/geburten-todesfaelle/geburten.html